CLINICAL TRIAL: NCT06702878
Title: A Group-Randomized, Standard-of-Care-Controlled, Crossover Trial Evaluating Nasal Antimicrobial Photodisinfection for the Prevention of Surgical Site Infections
Brief Title: Light-Activated Antimicrobial Therapy to Prevent Surgical Site Infections
Acronym: LANTERN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ondine Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: OBI-NPDT-SSI-004
Record Dates: First submitted 2024-11-12; First posted 2024-11-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Surgical Site Infections; Surgical Wound Infection; Infections; Anti-Infective Agents
Keywords: Surgical site infection; nasal decolonization; photodisinfection; nasal photodisinfection; Staphylococcus aureus; Photodynamic therapy; Methylene Blue; chlorhexidine; Disinfection
MeSH Terms: conditions — Surgical Wound Infection; Infections; Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: This study employs a group-randomized crossover design, comparing outcomes from the treatment group with that of a standard-of-care control group from the same hospitals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Nasal antimicrobial photodisinfection therapy (aPDT) (Experimental): Nasal antimicrobial photodisinfection therapy
  Interventions: Combination Product: nasal antimicrobial photodisinfection therapy
- Standard of Care Surgical Preventions - Control (No Intervention): Standard of Care surgical site prevention measures

INTERVENTIONS:
Combination Product: nasal antimicrobial photodisinfection therapy — Application of NF-031 solution (methylene blue 0.01% USP (methylthioninium chloride) and 0.25% chlorhexidine gluconate) in the nares followed by 2-minutes of light with nasal illuminators. The application is repeated a second time for total treatment time of 5-minutes.
  Arms: Nasal antimicrobial photodisinfection therapy (aPDT)

SUMMARY:
This is a Phase 3 multi-center, group-randomized, crossover trial to compare nasal antimicrobial photodisinfection therapy (aPDT) with standard of care for prevention of surgical site infections in patients undergoing major elective, urgent, or emergent surgeries in a hospital setting. The main outcomes are to:

1. compare the efficacy, and
2. estimate the safety of applying nasal (aPDT) before surgery in reducing the incidence of SSIs within the initial 30 days after surgery compared to standard of care (SOC).

Participants in the intervention group will receive aPDT prior to surgery on the day of surgery.

Participants in the control group will receive standard of care surgical site prevention measures prior to surgery.

DETAILED DESCRIPTION:
This study employs a group-randomized crossover design, comparing outcomes from the treatment group with that of a standard-of-care control group from the same hospitals. Each hospital ('site') engaged in the study will be randomly assigned to treatment plus standard-of-care or standard-of-care control on a 1:1 basis and will enroll patients into those respective groups during the first period of the study. After an approximate 6-week inactive interval period, each site will crossover to enroll the alternate group, up to a number of patients that matches the site's first period (or up to 10% more).

Eligible patients who successfully complete all screening assessments and meet inclusion and exclusion criteria will be enrolled. Patients in the treatment group will undergo aPDT treatment after admission to the preoperative area. All patients will be followed up for a 30-day post-surgery period. A patient-reported outcome (PRO) assessment to gauge the tolerability of the intervention after administration will also be performed in the treatment group.

Standard-of-care infection control practices will be applied according to infection prevention policies and procedures in place at each hospital. These practices are to remain unchanged for both groups throughout the study.

Microbiological samples will also be collected from any SSI and evaluated to establish the causative organism and its antibiotic susceptibility.

The incidence of SSIs during the 30-day postoperative period will be tracked to ensure comprehensive follow-up evaluations. In-person unscheduled visits will be conducted for medical assessment of suspected SSIs and collection of wound cultures.

Nasal Microbiota Substudy Approximately 500 study patients will have pre-treatment and post-treatment nasal swabs (in the treatment group) or single pre-surgical nasal swabs (in the control group) collected and stored. These samples will be processed for quantitative microbiological evaluation of S. aureus.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical patients, willing to sign the informed consent form and participate in the study.
2. ≥ 18 years of age
3. Presenting to an acute care hospital for major elective, urgent, or emergency surgery, defined as an open procedure involving a significant skin incision, including but not limited to the following types:

   1. Cardiac
   2. Vascular
   3. Orthopedic, including spine and 'clean' trauma
   4. Neurosurgery
   5. Breast surgeries
4. Are able to follow instructions, comply with protocol requirements, and participate in all required study visits.

Exclusion Criteria:

1. Pregnancy (current) or currently lactating. If patient is unsure of pregnancy status, a negative urine or serum pregnancy test (sensitive to 25 IU hCG) should be obtained within 14 days prior to surgery.
2. Surgical indication of infection.
3. History of surgery within 90 days prior to enrollment.
4. Anticipated surgery other than the index surgical procedure prior to patient's completion of the study.
5. Use of other nasal decolonization procedures on the day of surgery prior to the index procedure (mupirocin, povidone iodine, alcohol, etc.).
6. Patient has any medical, social or psychiatric condition(s) or current substance abuse condition that, in the opinion of the investigator, would preclude the patient's ability to provide informed consent, or to comply with the study requirements.
7. Enrollment in concomitant investigational research study in the past 30 days.

   Exclusion Criteria Specific to Treatment Group Patients Only:
8. Inability to tolerate insertion of the nasal light illuminator due to nasal obstructions or nares size, shape, or anatomical variants.
9. Known allergic reactions to components of the nasal disinfection treatment including methylene blue or chlorhexidine gluconate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4514 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Surgical Site Infection (SSI) within 30 days post surgery | Through 30 days post surgery
Percentage of Participants with Treatment-Related Adverse Events within 30 days after surgery. | Through 30 days post surgery

SECONDARY OUTCOMES:
Mean hospital length of stay after surgery | From day of surgery (from 1 day up to 30 days)
Number of hospital readmissions within 30 days of surgery | From day of surgery through 30 days post surgery
Number of Participants with Staph aureus nasal colonization following aPDT (substudy) | Immediately following aPDT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Simon Sinclair, MD, PhD, Study Director — Ondine Biomedical
Locations (16):
- United States (16):
  - Swedish Medical Center, Englewood, Colorado
  - HCA Brandon Florida, Brandon, Florida
  - HCA Florida Largo Hospital, Largo, Florida
  - HCA Florida NorthSide Hospital, St. Petersburg, Florida
  - HCA Florida Trinity Hospital, Trinity, Florida
  - Centennial Medical Center, Nashville, Tennessee
  - Medical City Dallas, Dallas, Texas
  - Medical City Heart and Spine Hospital, Dallas, Texas
  - Medical City Frisco Hospital, Frisco, Texas
  - HCA Houston Healthcare Kingwood, Kingwood, Texas
  - Medical City Plano, Plano, Texas
  - Methodist Metropolitan Hospital, San Antonio, Texas
  - Methodist Main Hospital and Landmark, San Antonio, Texas
  - Methodist Stone Oak, San Antonio, Texas
  - HCA Houston Healthcare Clear Lake Hospital, Webster, Texas
  - Johnston Willis Hospital, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No